CLINICAL TRIAL: NCT00204945
Title: Acute Responses in Diastolic Heart Failure
Brief Title: Catheterization Laboratory Study: Acute Responses in Diastolic Heart Failure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Wisconsin, Madison (Other)
Collaborators: Scios, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Health Services Research
Other Study IDs: 2001-496; K23 AGO01022
Record Dates: First submitted 2005-09-13; First posted 2005-09-20 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2019-02

CONDITIONS: Heart Failure, Congestive
Keywords: arterial stiffness; echocardiography; nesiritide; high heart pressures; cardiac catheterization
MeSH Terms: conditions — Heart Failure | interventions — Natriuretic Peptide, Brain

INTERVENTIONS:
Drug: nesiritide — a bolus, then infusion of nesiritide for 10-15 minutes

SUMMARY:
1. Research question: What is the response of the heart's pumping function to changes in heart chamber pressures?
2. Experimental design: Patients undergoing routine cardiac catheterization will be studied. A thermodilution pulmonary artery catheter will be inserted through a venous sheath and threaded into the pulmonary artery. After several minutes of quiet rest, baseline hemodynamics will be obtained, including a determination of cardiac output using thermodilution techniques and 30 seconds of pressure recordings from the left ventricle and proximal aorta. In addition, a brief echocardiogram will be performed, to determine ejection fraction and indices of diastolic filling. Finally, arterial tonometry will be obtained in quick succession from the brachial, radial, femoral, and carotid arteries. Following the collection of baseline data, a bolus and infusion of nesiritide will be started. After 10 minutes of nesiritide infusion, with the drug still infusing, a full set of invasive hemodynamics will again be obtained, as well as brief echocardiographic and arterial tonometry examinations.

ELIGIBILITY:
Inclusion Criteria:

* Cardiac catheterization

Exclusion Criteria:

* Unstable coronary syndrome,
* Critical coronary stenoses (>90%),
* Severe peripheral vascular disease,
* Symptomatic hypotension at completion of routine diagnostic cath,
* Significant valvular disease, resting heart rate >120 beats/min,
* Ejection fraction <45%,
* Presence of contraindications to nesiritide administration,
* Any evidence of clinical instability.

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 15 (Actual)
Dates: Start 2005-02; Primary Completion 2007-06-20 (Actual); Study Completion 2007-06-20 (Actual)

PRIMARY OUTCOMES:
arterial tonometry | following catheterization, then following 10 minutes of nesiritide infusion

CONTACTS AND LOCATIONS:
Overall Officials: Nancy K Sweitzer, MD PhD, Principal Investigator — University of Wisconsin, Madison
Locations (1):
- University of Wisconsin Hospital and Clinics, Madison, Wisconsin, United States